CLINICAL TRIAL: NCT02227719
Title: The Use of Customized Titanium Membrane for Horizontal Ridge Augmentation With Simultaneous Implant Placement
Brief Title: Customized Titanium Membrane for Growing Jaw Bone Horizontally
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hsun-Liang Chan, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00077102
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Bone Gain
Keywords: after augmentation; procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test: CTI (Experimental): CTI is titanium mesh
  Interventions: Device: CTI
- Control: Collagen membrane (Active Comparator): Collagen membrane is used for ridge augmentation
  Interventions: Device: Collagen membrane

INTERVENTIONS:
Device: CTI — CTI is the titanium mesh
  Arms: Test: CTI
Device: Collagen membrane
  Arms: Control: Collagen membrane

SUMMARY:
A single center, randomized, controlled, parallel-arm study is planned to investigate clinical outcomes of horizontal ridge augmentation with simultaneous single implant placement, using the newly designed Ti-membrane. Twenty-four adult subjects who fulfill the inclusion criteria will be enrolled. They will be randomly placed into one of two treatment groups: the customized titanium membrane (Cti-mem) or the collagen membrane (CM) group as a control. The decision of which material to use will be made after an implant is placed. Primary closure of the surgical site will be attempted for 4 months (+/- 1 month), after which the implants will be surgically uncovered and restored. Outcome analyses will be performed until 1-year after the crown will be placed, or 18 months (- 1 or +4 months) from the implant surgery. Clinical and radiographic parameters will be compared between the two experimental groups. The primary outcome is linear increase of horizontal ridge width from direct measurements.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age >18
* Overall good, stable health
* A single missing mandibular 1st molar for at least 3 months

Exclusion Criteria:

* Any medical conditions that may contradict implant and bone surgery or influence the outcome (detailed criteria in case report form)
* Pregnancy or lactating mothers
* Current heavy smokers (>10 cigarettes/day) or previous heavy smokers who have quit less than one year
* Unstable or unsuitable oral conditions for implant and bone surgery (detailed criteria in case report form)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
linear bone gain | 4 months after surgery

SECONDARY OUTCOMES:
implant marginal bone level | 18 months after baseline surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States